CLINICAL TRIAL: NCT04436562
Title: Phase 1 Open-label Study of the Absorption, Metabolism, and Excretion of Poziotinib Following a Single Oral Dose of [14C]-Poziotinib in Healthy Male Subjects
Brief Title: Study of the Absorption, Metabolism, and Excretion Following a Single Dose of [14C]-Poziotinib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPI-POZ-105
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Poziotinib (Experimental): A single oral dose of 8 mg poziotinib as a capsule formulation (as the hydrochloride salt) containing approximately 100 μCi of [14C]-poziotinib
  Interventions: Drug: [14C]-Poziotinib

INTERVENTIONS:
Drug: [14C]-Poziotinib — Single oral administration of 8 mg (as the hydrocholoride salt) of [14C]-poziotinib

SUMMARY:
This will be a Phase 1, open-label, nonrandomized, single-dose study in healthy male subjects to evaluate the Absorption, Metabolism, and Excretion of Poziotinib following a single oral dose of [14C]-poziotinib to healthy male subjects.

DETAILED DESCRIPTION:
Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Subjects will be admitted into the Clinical Research Unit (CRU) on Day -1. On the morning of Day 1, all subjects will receive a single oral dose of 8 mg (as the hydrochloride salt) containing approximately 100 μCi of [14C]-poziotinib in the fasted state.

Subjects will be confined to the CRU until at least Day 8.

Subjects will be discharged from the CRU on Day 8 if the following criteria are met:

* ≥90% mass balance recovery in combined urine and feces, and
* ≤1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 2 consecutive 24-hour periods in which fecal and urine samples are obtained.

If these criteria are not met by Day 8, subjects will remain in the CRU until all discharge criteria are met up to a maximum of Day 15 in order to continue 24-hour blood, urine, and feces collections, unless otherwise agreed upon by the Sponsor and Investigator.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2, inclusive
* In good health at Screening and/or at Check-in
* Subjects must be surgically sterile for at least 90 days, or when sexually active with female partners of childbearing and non-childbearing potential will be required to use a male condom with spermicide from CRU Check-in until 90 days after discharge. Subjects are required to refrain from donation of sperm from CRU Check-in until 90 days after discharge
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions
* History of at least 1 bowel movement per day

Key Exclusion Criteria:

* Stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Swallowing difficulties or ongoing diarrhea of any etiology
* Participation in a clinical study involving an investigational drug in the past 30 days prior to dosing
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in
* Use or intend to use any prescription medications/products within 14 days prior to Check-in
* Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in
* Exposure to significant diagnostic or therapeutic radiation or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
Cmax of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Time to Attain Maximum Observed Plasma Concentration (Tmax) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
Tmax of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC[last]) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
AUC(last) of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
AUC(inf) of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Percentage of AUCinf Derived by Extrapolation (%AUCext) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
%AUCext of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Apparent Terminal Elimination Half-Life (t1/2) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
t1/2 of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Elimination Rate Constant (λz, or kel) of [14C]-Poziotinib, Metabolites M1 and M2 | 1-15 days
λz, or kel of Total Radioactivity of [14C]-Poziotinib in Whole Blood and Plasma | 1-15 days
Apparent Volume of Distribution (VZ/F) During Terminal Phase of [14C]-Poziotinib | 1-15 days
Apparent Oral Clearance (CL/F) of [14C]-Poziotinib | 1-15 days
Whole Blood : Plasma Concentration Ratios of Total Radioactivity of [14C]-Poziotinib | 1-15 days
Total Radioactivity of Cumulative Amount Excreted in Urine (Aeu) | 1-15 days
Total Radioactivity of Fraction of Dose Excreted in Urine (feu) | 1-15 days
Total Radioactivity of Cumulative Amount Excreted in Feces (Aef) | 1-15 days
Total Radioactivity of Fraction of Dose Excreted in Feces (fef) | 1-15 days
Total Radioactivity of Cumulative Total Amount Excreted (Aetotal) | 1-15 days
Total Radioactivity of Fraction of Dose Excreted in Urine and Feces (fetotal) | 1-15 days
Poziotinib Metabolite Profiling and Identification in Plasma | 1-15 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | 1-15 days
Number of Participants with Hematology, Clinical Chemistry, Urinalysis Laboratory Abnormalities | 1-15 days
Number of Participants with 12-lead electrocardiograms (ECG) Abnormalities | 1-15 days
Number of Participants with Vital Sign and Physical Examinations Abnormalities | 1-15 days

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No